CLINICAL TRIAL: NCT00403078
Title: Stenting and Angioplasty With Protection in Patients At High-Risk for Endarterectomy (SAPPHIRE Worldwide)
Brief Title: SAPPHIRE Worldwide: Stenting and Angioplasty With Protection in Patients At High-Risk for Endarterectomy
Status: Completed | Type: Observational
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Sponsor
Other Study IDs: P06-3603
Record Dates: First submitted 2006-11-20; First posted 2006-11-23 (Estimated); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Carotid Artery Disease
Keywords: Carotid Artery Stenting (Endovascular)
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary objective of this study is to assess the outcomes of stenting with distal protection in the treatment of obstructive carotid artery disease. The devices to be utilized are the Cordis PRECISE® Nitinol Stent Systems (5.5F and 6F) and the Cordis ANGIOGUARD™ XP Emboli Capture Guidewire (ECGW).

DETAILED DESCRIPTION:
Carotid Artery Stenting

ELIGIBILITY:
Inclusion Criteria:

* High-surgical risk patients to be treated consistent with IFU labeling
* The patient or legally authorized representative has signed a written informed consent and HIPAA authorization, prior to the procedure, using a form that is approved by the Institutional Review Board or Medical Ethics Committee.

Exclusion Criteria:

* Patients not treated per the IFU
* Patients who are contraindicated per the IFU
* Patients previously enrolled in the study
* Patients requiring stenting of in-stent restenosis after CAS
* Inability or refusal to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will consist of high-surgical risk patients with atherosclerotic disease of the carotid artery(ies) from up to 350 clinical sites in the US and Canada.
Sampling Method: Non-Probability Sample
Enrollment: 21008 (Actual)
Dates: Start 2006-10; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Any death, stroke or any MI | up to 30-days post-procedure

SECONDARY OUTCOMES:
Assess the consistency of MAE rates of stenting with distal protection in the treatment of obstructive carotid artery disease among high, medium and low volume centers with physicians who have validated CASES training levels of 1, 2, 2P or 3 | 30 days
Assess the real-world cost-effectiveness of carotid artery stenting in subjects enrolled | Every follow-up where a PRO instrument QoL was assessed
Estimate MAE (death and ipsilateral stroke) rate in a subset of the planned total enrollment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Dave, MD, Principal Investigator — Harrisburg Hospital, 2808 Old Post Rd., Harrisburg, PA 17110; Robert Hibbard, MD, Principal Investigator — Bryan LGH Heart Institute, 1500 South 48th St, Suite 400, Lincoln, NE 68506; Douglas Massop, MD, Principal Investigator — Iowa Clinic-Heart and Vascular Care, 5950 University Ave, West Des Moines, IA 50266; Christopher Metzger, MD, Principal Investigator — The Heart Center, PC, 2050 Meadowview Parkway, Kingsport, TN 37660
Locations (5):
- United States (5):
  - Christiana Care Health Services, Newark, Delaware
  - Iowa Clinic, Heart & Vascular Care, West Des Moines, Iowa
  - Bryan LGH Heart Institute, Lincoln, Nebraska
  - Harrisburg Hospital, Harrisburg, Pennsylvania
  - The Heart Center, PC, Kingsport, Tennessee

REFERENCES:
- [Result] Massop D, Dave R, Metzger C, Bachinsky W, Solis M, Shah R, Schultz G, Schreiber T, Ashchi M, Hibbard R; SAPPHIRE Worldwide Investigators. Stenting and angioplasty with protection in patients at high-risk for endarterectomy: SAPPHIRE Worldwide Registry first 2,001 patients. Catheter Cardiovasc Interv. 2009 Feb 1;73(2):129-36. doi: 10.1002/ccd.21844. PMID 18924164
- [Derived] Qureshi O, Mena-Hurtado C, Romain G, Cleman J, Callegari S, Smolderen KG. Applying a Random Forest Approach in Predicting Health Status in Patients with Carotid Artery Stenosis 30 Days Post Stenting. Stroke Vasc Interv Neurol. 2025 Sep 26;5(6):e001938. doi: 10.1161/SVIN.125.001938. eCollection 2025 Nov. PMID 41608717